CLINICAL TRIAL: NCT06500559
Title: Comparison of Alveolar Bone Dehiscence and Fenestration Following Maxillary Canine Retraction Using Two Methods of Tooth Movement Acceleration. A Randomized Clinical Trial
Brief Title: Alveolar Bone Dehiscence and Fenestration Following Accelerated Maxillary Canine Retraction
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tanta University (Other)
Responsible Party: Principal Investigator, Safa Basiouny Alawy, Lecturer of Orthodontics, Tanta University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: #R-ORTH-6-24-3117
Record Dates: First submitted 2024-07-08; First posted 2024-07-15 (Actual); Last update posted 2025-09-10 (Actual); Status verified 2025-09

CONDITIONS: Fenestration; Dehiscence
Keywords: accelerated orthodontics; Dehiscence; fenestration; CBCT

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- group I: PRP injection (Experimental): Accelerated maxillary canine retraction will be done after PRP injection in one random side of the maxillary arch while the other side serve as control
  Interventions: Procedure: PRP injection
- group II: Combined decortication and PRP injection (Experimental): Accelerated maxillary canine retraction will be done after combined decortication and PRP injection in one random side of the maxillary arch while the other side serve as control
  Interventions: Procedure: Combined decortication and PRP injection

INTERVENTIONS:
Procedure: PRP injection — PRP (0.7 ml = 70 unit) will be injected submucosal disto-buccal and disto-palatal to the maxillary canine like the local anesthesia injection in group I experimental sides
  Arms: group I: PRP injection
Procedure: Combined decortication and PRP injection — Experimental sides will receive PRP injection after performing decortication. After administration of local anesthesia, two-line flap will be performed from the mesial surface of the maxillary second premolar to the distal surface of the maxillary canine Mucoperiosteal flap will be reflected in the buccal side. Two millimeters of marginal crestal bone will be held intact and using a high-speed drill and a round carbide bur (1mm diameter) under copious saline irrigation, the cortical wall will be penetrated to reach marrow spaces. Multiple perforations (10 holes for standardization) in the cortical bone will be created. The surgical site will then rinsed, and the flap will be repositioned and sutured.
  Arms: group II: Combined decortication and PRP injection

SUMMARY:
Alveolar bone loss and fenestration are the most prevalent bone defects that often result in root exposure, gingival recession, and potential treatment relapse or failure. These issues present complications in orthodontic therapy. Hence, reducing the length of orthodontic therapy and minimizing the occurrence of these serious complications are highly important for orthodontic patients, particularly adults. platelet-rich plasma (PRP) injection and decortication are two promising methods for accelerated tooth movements. Thus, The aim of this study is to evaluate alveolar bone dehiscence and fenestrations after canine retraction, using alveolar decortication and PRP injection as two methods for accelerating tooth movements.

ELIGIBILITY:
Inclusion Criteria:

1. Age of the patients ranged from 16: 22 years old.
2. Malocclusion that requires extraction of the maxillary first premolar and canine retraction (e.g. class I bimaxillary dentoalveolar protrusion and class II div 1 malocclusion).
3. Maximum anchorage needed for the maxillary arch as a part of the orthodontic treatment plan.
4. Good oral hygiene and periodontal condition.

Exclusion Criteria:

1. Medically compromised patients.
2. Severe crowding in the maxillary arch.
3. Chronic intake of NSAIDs or any medication that interfere with OTM.
4. Previous orthodontic treatment.

Ages: 16 Years to 22 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 60 (Actual)
Dates: Start 2024-05-01 (Actual); Primary Completion 2025-02-01 (Actual); Study Completion 2025-09-07 (Actual)

PRIMARY OUTCOMES:
Alveolar bone dehiscence | 4 months
  Pre- and post- retraction CBCTs will be obtained from patients. Linear measurement (mm) for dehiscence (LM-D) will be defined as the distance between the alveolar crest to the cementoenamel junction of each root (critical point will be set at 2 mm)
Alveolar bone fenestration | 4 months
  Pre- and post- retraction CBCTs will be obtained from patients. Linear measurement (mm) for fenestration (LM-F) will be recorded when the defect involved only the apical one-third of a root (critical point will be set at 2.2 mm)

CONTACTS AND LOCATIONS:
Locations (1):
- Tanta University, Tanta, Tanta, Egypt

IPD SHARING:
Plan to Share IPD: No